CLINICAL TRIAL: NCT03731429
Title: Efficiency of Intravenous Lidocaine to Reduce Coughing and the Hemodynamic Changes Associated to Tracheal Extubation
Brief Title: Lidocaine to Prevent Cough and Hemodynamic Changes in Tracheal Extubation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Fernandez (Other)
Responsible Party: Principal Investigator, Santiago Ficcadenti, Principal investigator, Hospital Fernandez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201824
Record Dates: First submitted 2018-10-22; First posted 2018-11-06 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Lidocaine
Keywords: Cough; Sore throat; Hemodynamic changes; Extubation; Lidocaine; Double blind
MeSH Terms: conditions — Cough; Pharyngitis | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study was designed as a double-blind randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Group that receives a 1 mg/kg single bolus of 2% IV lidocaine
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): group that receives 0.9% saline solution
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Lidocaine — prior to extubation
  Other Names: GOBBI
  Arms: Intervention
Drug: Saline Solution — Prior to extubation
  Other Names: GOBBI
  Arms: Placebo

SUMMARY:
Coughing during tracheal extubation can be associated to adverse effects like tachycardia, arterial hypertension (AHT), increase of intracranial pressure (ICP) and intraocular pressure (IOP), and the dehiscence of surgical wounds. In ophthalmic, head and neck, and abdominal surgery, and in several other neurosurgical interventions it is vital to prevent these effects. The incidence of laryngeal irritation due to orotracheal intubation hinders patient comfort in the immediate postoperative (POP) period and no pharmacological intervention has been yet proven to prevent it.

At the end of the surgical procedure, the depth of the anesthetic plane decreases with the concomitant suspension of the anesthetic agents. However, the patient still requires ventilatory support through the endotracheal tube (EDT). The physical stimulation of the trachea created by this foreign body leads to the activation of the sympathetic nervous system, expressed in AHT, tachycardia, and ICP. To tolerate the EDT and prevent these effects, different maneuvers have been tested such as extubating the patient in a deep anesthetic plane or administering intravenous (IV) narcotics with the entailed complications: airway (AW) obstruction and hypercapnia, and the aspiration of an unprotected AW. Progress has been made with the introduction of ultrashort acting opioids, with significant statistical results. Moreover, beta-blockers, calcium channel blockers, angiotensin converting enzyme inhibitors and dexmedetomidine have been used to decrease the hemodynamic impact associated to tracheal extubation. The use of both IV and intratracheal lidocaine in doses ranging from 1 mg/kg to 3 mg/kg, has been studied with controversial results.

In view of the above, and as lidocaine is the most commonly used low-cost drug in all operating rooms with a good safety profile when used at low doses, the purpose of this study is twofold: to assess its effects at reducing coughing and to evaluate its hemodynamic impact when administering IV 1 mg/kg prior to extubation. Then, the efficiency of reducing the incidence of sore throats after the immediate POP shall be investigated.

ELIGIBILITY:
Inclusion criteria:

* American Society of Anesthesiologists Risk I & II.
* Age 18-65 years.
* Scheduled for: cholecystectomy, hernioplasty or laparoscopic gynecological surgery, under balanced general anesthesia (GA) and orotracheal intubation (OTI).

Exclusion criteria:

* Local anesthetic (LA) allergy.
* Presence of predictors of potentially difficult intubation (DI) according to criteria defined by the American Society of Anesthesiologists.
* Upper airway inflammatory symptoms during the previous week.
* Chronic kidney disease with clearance lower than 60 ml/m using the Modification of Diet in Renal Disease (MDRD) equation.
* Child-Pugh B-C liver disease.
* Treated with ACEinhibitors and/or BB.
* Second and third grade atrioventricular block.
* Symptomatic bradycardia.
* Tachyarrhythmias.
* Left bundle branch block (LBBB).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-09-19 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Determine the efficiency of IV lidocaine in reducing the incidence of coughing | From the moment the endotracheal tube is retired to 5 minutes after
  Apply the Minogue scale to assess the coughing associated to tracheal extubation.
  Modified Minogue scale by Likert: (ordinal, 0 to 5)
  Grade 1: absence of coughing and muscle stiffness Grade 2: transient coughing while removing EDT Grade 3: moderate cough (3 or less coughing episodes each lasting one or two seconds) Grade 4: muscular stiffness or severe cough (4 ore more episodes lasting more tham two seconds) Grade 5: laryngospasm
Determine the efficiency of IV lidocaine in reducing the arterial hypertension associated with tracheal extubation | From the end of anesthesia to 5 minutes after tracheal extubation (At time 0, time 2 and time 3)
  Gather mean arterial pressure (MAP) record at the time of the extubation.
  Difference in MAP between anesthesia ceasing (time 0) and extubation (time 2) (continuous, mmHg) Difference in MAP between time 0 and 5 minutes after extubation (time 3) (continuous, mmHg)
Determine the efficiency of IV lidocaine in reducing the increase in heart rate (HR) associated with tracheal extubation | From the end of anesthesia to 5 minutes after tracheal extubation (At time 0, time 2 and time 3)
  Gather HR record at the time of the extubation.
  Difference in HR between time 0 and time 2 (discreet, bpm) Difference in HR between time 0 and time 3 (discreet, bpm)

SECONDARY OUTCOMES:
Record the time elapsed from the end of anesthesia and the administration of lidocaine to extubation. | Intraoperative. From the end of anesthesia (time 0) to tracheal extubation (time 2)
  As a safety event. Record time between t0 and t2 (continuous, minutes)
Assess immediate POP sore throat | 30 minutes after extubation
  using the Likert ten-point severity pain scale. The scale ranges from 0 to 10. 0 equals no pain, and 10 indicates the worst pain.

OTHER OUTCOMES:
Monitor the adverse reactions (AR) that may occur after the administration of IV lidocaine and report them | 24 hours after extubation
  Severe and unexpected AR shall be reported according to Argentina's National Administration of Drugs, Food and Medical Technology (ANMAT) with the means appropriate and intended for that purpose. Likewise, this scenario will be immediately reported to the Fernández hospital Ethics and Research Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Ficcadenti, Doctor, Principal Investigator — Hospital Fernandez
Locations (1):
- Hospital Fernandez, Capital Federal, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Minogue SC, Ralph J, Lampa MJ. Laryngotracheal topicalization with lidocaine before intubation decreases the incidence of coughing on emergence from general anesthesia. Anesth Analg. 2004 Oct;99(4):1253-1257. doi: 10.1213/01.ANE.0000132779.27085.52. PMID 15385385
- [Result] Hohlrieder M, Tiefenthaler W, Klaus H, Gabl M, Kavakebi P, Keller C, Benzer A. Effect of total intravenous anaesthesia and balanced anaesthesia on the frequency of coughing during emergence from the anaesthesia. Br J Anaesth. 2007 Oct;99(4):587-91. doi: 10.1093/bja/aem203. Epub 2007 Jul 27. PMID 17660457
- [Result] Bruder N, Pellissier D, Grillot P, Gouin F. Cerebral hyperemia during recovery from general anesthesia in neurosurgical patients. Anesth Analg. 2002 Mar;94(3):650-4; table of contents. doi: 10.1097/00000539-200203000-00031. PMID 11867391
- [Result] Coles JP, Leary TS, Monteiro JN, Brazier P, Summors A, Doyle P, Matta BF, Gupta AK. Propofol anesthesia for craniotomy: a double-blind comparison of remifentanil, alfentanil, and fentanyl. J Neurosurg Anesthesiol. 2000 Jan;12(1):15-20. doi: 10.1097/00008506-200001000-00004. PMID 10636615
- [Result] Talke P, Caldwell JE, Brown R, Dodson B, Howley J, Richardson CA. A comparison of three anesthetic techniques in patients undergoing craniotomy for supratentorial intracranial surgery. Anesth Analg. 2002 Aug;95(2):430-5, table of contents. doi: 10.1097/00000539-200208000-00036. PMID 12145066
- [Result] Christensen AM, Willemoes-Larsen H, Lundby L, Jakobsen KB. Postoperative throat complaints after tracheal intubation. Br J Anaesth. 1994 Dec;73(6):786-7. doi: 10.1093/bja/73.6.786. PMID 7880666
- [Result] Harding CJ, McVey FK. Interview method affects incidence of postoperative sore throat. Anaesthesia. 1987 Oct;42(10):1104-7. doi: 10.1111/j.1365-2044.1987.tb05179.x. PMID 3688395
- [Result] Herlevsen P, Bredahl C, Hindsholm K, Kruhoffer PK. Prophylactic laryngo-tracheal aerosolized lidocaine against postoperative sore throat. Acta Anaesthesiol Scand. 1992 Aug;36(6):505-7. doi: 10.1111/j.1399-6576.1992.tb03507.x. PMID 1514331
- [Result] Lee B, Lee JR, Na S. Targeting smooth emergence: the effect site concentration of remifentanil for preventing cough during emergence during propofol-remifentanil anaesthesia for thyroid surgery. Br J Anaesth. 2009 Jun;102(6):775-8. doi: 10.1093/bja/aep090. Epub 2009 May 2. PMID 19411668
- [Result] Mayhan WG. Disruption of blood-brain barrier during acute hypertension in adult and aged rats. Am J Physiol. 1990 Jun;258(6 Pt 2):H1735-8. doi: 10.1152/ajpheart.1990.258.6.H1735. PMID 2113773
- [Result] Gauthier A, Girard F, Boudreault D, Ruel M, Todorov A. Sevoflurane provides faster recovery and postoperative neurological assessment than isoflurane in long-duration neurosurgical cases. Anesth Analg. 2002 Nov;95(5):1384-8, table of contents. doi: 10.1097/00000539-200211000-00052. PMID 12401630
- [Result] Lowrie A, Johnston PL, Fell D, Robinson SL. Cardiovascular and plasma catecholamine responses at tracheal extubation. Br J Anaesth. 1992 Mar;68(3):261-3. doi: 10.1093/bja/68.3.261. PMID 1547048
- [Result] Grillo P, Bruder N, Auquier P, Pellissier D, Gouin F. Esmolol blunts the cerebral blood flow velocity increase during emergence from anesthesia in neurosurgical patients. Anesth Analg. 2003 Apr;96(4):1145-1149. doi: 10.1213/01.ANE.0000055647.54957.77. PMID 12651674
- [Result] Muzzi DA, Black S, Losasso TJ, Cucchiara RF. Labetalol and esmolol in the control of hypertension after intracranial surgery. Anesth Analg. 1990 Jan;70(1):68-71. PMID 1967515
- [Result] Fujii Y, Saitoh Y, Takahashi S, Toyooka H. Combined diltiazem and lidocaine reduces cardiovascular responses to tracheal extubation and anesthesia emergence in hypertensive patients. Can J Anaesth. 1999 Oct;46(10):952-6. doi: 10.1007/BF03013130. PMID 10522582 (Retraction: PMID 23625550 Can J Anaesth. 2013 Jun;60(6):613)
- [Result] Tsutsui T. Combined administration of diltiazem and nicardipine attenuates hypertensive responses to emergence and extubation. J Neurosurg Anesthesiol. 2002 Apr;14(2):89-95. doi: 10.1097/00008506-200204000-00001. PMID 11907387
- [Result] Kross RA, Ferri E, Leung D, Pratila M, Broad C, Veronesi M, Melendez JA. A comparative study between a calcium channel blocker (Nicardipine) and a combined alpha-beta-blocker (Labetalol) for the control of emergence hypertension during craniotomy for tumor surgery. Anesth Analg. 2000 Oct;91(4):904-9. doi: 10.1097/00000539-200010000-00024. PMID 11004045
- [Result] Tanskanen PE, Kytta JV, Randell TT, Aantaa RE. Dexmedetomidine as an anaesthetic adjuvant in patients undergoing intracranial tumour surgery: a double-blind, randomized and placebo-controlled study. Br J Anaesth. 2006 Nov;97(5):658-65. doi: 10.1093/bja/ael220. Epub 2006 Aug 16. PMID 16914460
- [Result] Nho JS, Lee SY, Kang JM, Kim MC, Choi YK, Shin OY, Kim DS, Kwon MI. Effects of maintaining a remifentanil infusion on the recovery profiles during emergence from anaesthesia and tracheal extubation. Br J Anaesth. 2009 Dec;103(6):817-21. doi: 10.1093/bja/aep307. Epub 2009 Oct 28. PMID 19864308
- [Result] Shajar MA, Thompson JP, Hall AP, Leslie NA, Fox AJ. Effect of a remifentanil bolus dose on the cardiovascular response to emergence from anaesthesia and tracheal extubation. Br J Anaesth. 1999 Oct;83(4):654-6. doi: 10.1093/bja/83.4.654. PMID 10673886
- [Result] Ghodraty MR, Hasani V, Bagheri-Aghdam A, Zamani MM, Pournajafian A, Rokhtabnak F, Kholdebarin A, Nader ND. Remifentanil infusion during emergence moderates hemodynamic and cough responses to the tracheal tube: A randomized controlled trial. J Clin Anesth. 2016 Sep;33:514-20. doi: 10.1016/j.jclinane.2015.09.001. Epub 2015 Oct 23. PMID 26603110
- [Result] Altintas F, Bozkurt P, Kaya G, Akkan G. Lidocaine 10% in the endotracheal tube cuff: blood concentrations, haemodynamic and clinical effects. Eur J Anaesthesiol. 2000 Jul;17(7):436-42. doi: 10.1046/j.1365-2346.2000.00696.x. PMID 10964145
- [Result] Prengel AW, Lindner KH, Hahnel JH, Georgieff M. Pharmacokinetics and technique of endotracheal and deep endobronchial lidocaine administration. Anesth Analg. 1993 Nov;77(5):985-9. doi: 10.1213/00000539-199311000-00019. PMID 8214738
- [Result] Baraka A. Intravenous lidocaine controls extubation laryngospasm in children. Anesth Analg. 1978 Jul-Aug;57(4):506-7. doi: 10.1213/00000539-197807000-00028. No abstract available. PMID 360878
- [Result] Bidwai AV, Bidwai VA, Rogers CR, Stanley TH. Blood-pressure and pulse-rate responses to endotracheal extubation with and without prior injection of lidocaine. Anesthesiology. 1979 Aug;51(2):171-3. doi: 10.1097/00000542-197908000-00020. No abstract available. PMID 453622
- [Result] Copeland SE, Ladd LA, Gu XQ, Mather LE. The effects of general anesthesia on whole body and regional pharmacokinetics of local anesthetics at toxic doses. Anesth Analg. 2008 May;106(5):1440-9, table of contents. doi: 10.1213/ane.0b013e31816ba541. PMID 18420858
- [Result] Copeland SE, Ladd LA, Gu XQ, Mather LE. The effects of general anesthesia on the central nervous and cardiovascular system toxicity of local anesthetics. Anesth Analg. 2008 May;106(5):1429-39, table of contents. doi: 10.1213/ane.0b013e31816d12af. PMID 18420857
- [Result] Shankar Ramaswamy, John A. Wilson, Lesley Colvin. Non-opioid-based adjuvant analgesia in perioperative care. Continuing Education in Anaesthesia, Critical Care & Pain. 2013; 13:152-7.
- [Result] N Eipe, S Gupta, J Penning. Intravenous lidocaine for acute pain: an evidence-based clinical update. Br J Anaesth Education. 2016; 16:292-8.
- [Result] Mazzone SB, Undem BJ. Cough sensors. V. Pharmacological modulation of cough sensors. Handb Exp Pharmacol. 2009;(187):99-127. doi: 10.1007/978-3-540-79842-2_6. PMID 18825338
- [Result] STEINHAUS JE, GASKIN L. A study of intravenous lidocaine as a suppressant of cough reflex. Anesthesiology. 1963 May-Jun;24:285-90. doi: 10.1097/00000542-196305000-00006. No abstract available. PMID 13983769
- [Result] Martínez-Zúñiga JP, Lorenzo-Balderas, Silva-Escobedo JG. Lidocaine in low doses combining intravenous and endotracheal therapies: reduces incidence of coughing and hemodynamic changes during extubation. Rev Sanid Milit Mex. 2011; 65:95-8.
- [Result] Zamora Lozano J, Cruz Villasenor JA, Rodriguez Reyes J, Sanchez Rodriguez JP, Briones Corona G, Gallardo Alonso LA. [Comparison of topical, intravenous, and intracuff lidocaine for reducing coughing after extubation during emergence from general anesthesia]. Rev Esp Anestesiol Reanim. 2007 Dec;54(10):596-601. Spanish. PMID 18200994
- [Result] Saghaei M, Reisinejad A, Soltani H. Prophylactic versus therapeutic administration of intravenous lidocaine for suppression of post-extubation cough following cataract surgery: a randomized double blind placebo controlled clinical trial. Acta Anaesthesiol Taiwan. 2005 Dec;43(4):205-9. PMID 16450594
- [Result] Lee JH, Koo BN, Jeong JJ, Kim HS, Lee JR. Differential effects of lidocaine and remifentanil on response to the tracheal tube during emergence from general anaesthesia. Br J Anaesth. 2011 Mar;106(3):410-5. doi: 10.1093/bja/aeq396. Epub 2011 Jan 2. PMID 21205628
- [Result] Williams KA, Barker GL, Harwood RJ, Woodall NM. Combined nebulization and spray-as-you-go topical local anaesthesia of the airway. Br J Anaesth. 2005 Oct;95(4):549-53. doi: 10.1093/bja/aei202. Epub 2005 Aug 26. PMID 16126785
- [Result] Mainland PA, Kong AS, Chung DC, Chan CH, Lai CK. Absorption of lidocaine during aspiration anesthesia of the airway. J Clin Anesth. 2001 Sep;13(6):440-6. doi: 10.1016/s0952-8180(01)00298-7. PMID 11578889
- [Result] Rosenberg PH, Veering BT, Urmey WF. Maximum recommended doses of local anesthetics: a multifactorial concept. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):564-75; discussion 524. doi: 10.1016/j.rapm.2004.08.003. PMID 15635516
- [Result] Donald MJ, Derbyshire S. Lignocaine toxicity; a complication of local anaesthesia administered in the community. Emerg Med J. 2004 Mar;21(2):249-50. doi: 10.1136/emj.2003.008730. PMID 14988367
- [Result] Scuderi PE. Postoperative sore throat: more answers than questions. Anesth Analg. 2010 Oct;111(4):831-2. doi: 10.1213/ANE.0b013e3181ee85c7. No abstract available. PMID 20870978
- [Result] Minto CF, Schnider TW, Egan TD, Youngs E, Lemmens HJ, Gambus PL, Billard V, Hoke JF, Moore KH, Hermann DJ, Muir KT, Mandema JW, Shafer SL. Influence of age and gender on the pharmacokinetics and pharmacodynamics of remifentanil. I. Model development. Anesthesiology. 1997 Jan;86(1):10-23. doi: 10.1097/00000542-199701000-00004. PMID 9009935
- [Result] Minto CF, Schnider TW, Shafer SL. Pharmacokinetics and pharmacodynamics of remifentanil. II. Model application. Anesthesiology. 1997 Jan;86(1):24-33. doi: 10.1097/00000542-199701000-00005. PMID 9009936
- [Result] Kapila A, Glass PS, Jacobs JR, Muir KT, Hermann DJ, Shiraishi M, Howell S, Smith RL. Measured context-sensitive half-times of remifentanil and alfentanil. Anesthesiology. 1995 Nov;83(5):968-75. doi: 10.1097/00000542-199511000-00009. PMID 7486182
- [Result] Burkle H, Dunbar S, Van Aken H. Remifentanil: a novel, short-acting, mu-opioid. Anesth Analg. 1996 Sep;83(3):646-51. doi: 10.1097/00000539-199609000-00038. PMID 8780298
- [Result] Egan TD, Lemmens HJ, Fiset P, Hermann DJ, Muir KT, Stanski DR, Shafer SL. The pharmacokinetics of the new short-acting opioid remifentanil (GI87084B) in healthy adult male volunteers. Anesthesiology. 1993 Nov;79(5):881-92. doi: 10.1097/00000542-199311000-00004. PMID 7902032
- [Result] Kim H, Min KT, Lee JR, Ha SH, Lee WK, Seo JH, Choi SH. Comparison of Dexmedetomidine and Remifentanil on Airway Reflex and Hemodynamic Changes during Recovery after Craniotomy. Yonsei Med J. 2016 Jul;57(4):980-6. doi: 10.3349/ymj.2016.57.4.980. PMID 27189295
- [Result] Ikeda Y, Oda Y, Nakamura T, Takahashi R, Miyake W, Hase I, Asada A. Pharmacokinetics of lidocaine, bupivacaine, and levobupivacaine in plasma and brain in awake rats. Anesthesiology. 2010 Jun;112(6):1396-403. doi: 10.1097/ALN.0b013e3181d9cc54. PMID 20460991